CLINICAL TRIAL: NCT02419534
Title: Randomized Controlled Trial Comparing the Efficacy of Polyethylene Glycol Alone and Polyethylene Glycol Combined With Topical Diltiazem in Treating Anal ﬁssure in Children
Brief Title: Pediatrics Anal Fissures Treatment With Polyethylene Glycol
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Ayman Aljazaeri, Assistant Professor & Consultant of Pediatric surgery, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14/4293
Record Dates: First submitted 2015-04-02; First posted 2015-04-17 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Fissure in Ano
Keywords: Pediatric, fissure in ano
MeSH Terms: conditions — Fissure in Ano | interventions — Polyethylene Glycols; Diltiazem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyethylene glycol (Active Comparator): In our study parents will be asked to start at 1g per day if they are less than 1 year of age and 2g per day in divided doses if they are older and will be asked to titrate the does according to the response up to the a maximum does of .5g/kg/day. In titrating the dose parent will be asked to increase the dose every 2 days until the child pass one normal BM per day without significant efforts. They should titrate down or hold treatment if the child developed lose BM or diarrhea. Caregiver will be asked to use placebo ointment by applying 5mm on fingertip to the anal verge area twice a day for the duration of the study.
  Interventions: Drug: Polyethylene glycol
- Polyethylene glycol with Diltiazem (Active Comparator): Parents will be instructed to apply 5 mm of ointment on a fingertip at the anal verge twice daily for the duration of the study
  Interventions: Drug: Polyethylene glycol with Diltiazem

INTERVENTIONS:
Drug: Polyethylene glycol — Laxative to treat constipation
  Other Names: Movicol
  Arms: Polyethylene glycol
Drug: Polyethylene glycol with Diltiazem — Laxative and topical calcium channel blocker
  Other Names: Movicol + Diltiazem
  Arms: Polyethylene glycol with Diltiazem

SUMMARY:
To evaluate whether effectively treating anal fissure-associated constipation using oral PEG alone can eliminate the inconvenience of add topical agent such as DTZ. As previous studies have shown the topical agent are more effective in treating anal fissure when combined with less effective laxatives

DETAILED DESCRIPTION:
Anal fissure (AF) is common among children attending pediatric and surgery clinics and is frequently associated with painful defecation, stool withholding and constipation which affect 1%-30% of the pediatric population. Constipated children consume low fiber diets, come from lower socioeconomic families and tend to be obese. The reason why anal fissure develops is still largely unclear, however the pathogenesis points to an initial anal trauma cause by the hard stool leading to anal sphincter hypertonia or spasm which cause local ischemia and non-healing ulcer. It is not clear why the posterior anal canal is the most affected part by the local anal ischemia.

Current medical therapy for chronic anal fissure focuses on alleviating the two main pathologies by using anal sphincter relaxing topical ointments and laxative to treat associated constipation. The classical text book described treatment of AF focus on increasing fiber intake to treat the underlying constipation. Jensen et al, has found that treating the first episode of anal fissure with bran is more effective than local anesthetic or steroids. The American Society of Colon and Rectal Surgeons practice parameters suggest that increase in fluid and fiber ingestion, use of sitz baths, and if necessary use of stool softeners are safe have few side effects and should be the initial therapy for all patients with anal fissure.

There have been many recent randomized trials describing the effectiveness of Nitroglycerin (NTG), Botulinum toxin injection or the topical calcium channel blockers such as Diltiazem (DTZ) in adult and pediatric. A systematic review of the available randomized trials of these agents has shown that topical agents are marginally better than placebo [15]. Furthermore, in most trials that have demonstrated the effectiveness of topical agents laxatives usage was either not well controlled or lactulose was the main agent used. In children, many recent randomized trials have demonstrated the superior effectiveness of PEG over lactulose consequently; we think that treating AF with PEG is likely to improve the success rate and lead to persistent log-term fissure healing. Most adults and pediatric RCTs that have demonstrated the effectiveness of topical agents in healing AF, have focused on comparing various topical agents to placebo in treating AF, however the effectiveness in comparison to placebo has never been demonstrated in patients how are placed on more effective laxative such as PEG. We hypothesize that replacing lactulose with a more effective laxative such PEG as a sole agent to treat AF can eliminate the effectiveness and therefore the need to add topical sphincter relaxing agent such DTZ or NTG. Laxative-only treatment is likely to be more convenient and more cost-effective.

ELIGIBILITY:
Inclusion Criteria:

1. Painful defecation with visible anal fissure
2. Symptoms for 2 weeks
3. Children less than 14 years of age

Exclusion Criteria:

1. Previous surgeries
2. Chronic illness affecting the rectum or perianal area
3. Refuse to participate

Ages: 1 Minute to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Number of cases with healed anal fissure as detected by clinical physical exam | up to 8 weeks

SECONDARY OUTCOMES:
Number cases with painless bowel movement detected during clinical visits or phone interviews | at 2,4 and 8 weeks
Number of individuals with minimal or no straining during bowel movement detected during clinical visits or phone interviews | at 2, 4, and 8 weeks
Number of cases that are passing soft bowel movements detected during clinical visits or phone interviews | at 2, 4, and 8 weeks
Number of cases who are passing > 3 watery bowel movement (Diarrhea) detected during clinical visits or phone interviews | at 2, 4, and 8 weeks
Compliance (number of cases who are taking the PEG and/or Diltiazem Ointment) as detected during clinical visits or phone interviews | 2, 4, and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Al-Jazaeri, Principal Investigator — Associate Professor & Consultant of Pediatric,Medical College, King Saud University
Locations (1):
- College of medicine, king saud university, Riyadh, Nejd Province - Central, Saudi Arabia

REFERENCES:
- [Result] Mugie SM, Benninga MA, Di Lorenzo C. Epidemiology of constipation in children and adults: a systematic review. Best Pract Res Clin Gastroenterol. 2011 Feb;25(1):3-18. doi: 10.1016/j.bpg.2010.12.010. PMID 21382575
- [Result] Sonmez K, Demirogullari B, Ekingen G, Turkyilmaz Z, Karabulut R, Basaklar AC, Kale N. Randomized, placebo-controlled treatment of anal fissure by lidocaine, EMLA, and GTN in children. J Pediatr Surg. 2002 Sep;37(9):1313-6. doi: 10.1053/jpsu.2002.34997. PMID 12194122
- [Result] Farouk R, Duthie GS, MacGregor AB, Bartolo DC. Sustained internal sphincter hypertonia in patients with chronic anal fissure. Dis Colon Rectum. 1994 May;37(5):424-9. doi: 10.1007/BF02076185. PMID 8181401
- [Result] Poh A, Tan KY, Seow-Choen F. Innovations in chronic anal fissure treatment: A systematic review. World J Gastrointest Surg. 2010 Jul 27;2(7):231-41. doi: 10.4240/wjgs.v2.i7.231. PMID 21160880
- [Result] Schouten WR, Briel JW, Auwerda JJ. Relationship between anal pressure and anodermal blood flow. The vascular pathogenesis of anal fissures. Dis Colon Rectum. 1994 Jul;37(7):664-9. doi: 10.1007/BF02054409. PMID 8026232
- [Result] Jensen SL. Treatment of first episodes of acute anal fissure: prospective randomised study of lignocaine ointment versus hydrocortisone ointment or warm sitz baths plus bran. Br Med J (Clin Res Ed). 1986 May 3;292(6529):1167-9. doi: 10.1136/bmj.292.6529.1167. PMID 3011180
- [Result] Perry WB, Dykes SL, Buie WD, Rafferty JF; Standards Practice Task Force of the American Society of Colon and Rectal Surgeons. Practice parameters for the management of anal fissures (3rd revision). Dis Colon Rectum. 2010 Aug;53(8):1110-5. doi: 10.1007/DCR.0b013e3181e23dfe. No abstract available. PMID 20628272
- [Result] Samim M, Twigt B, Stoker L, Pronk A. Topical diltiazem cream versus botulinum toxin a for the treatment of chronic anal fissure: a double-blind randomized clinical trial. Ann Surg. 2012 Jan;255(1):18-22. doi: 10.1097/SLA.0b013e318225178a. PMID 21685792
- [Result] Ala S, Saeedi M, Hadianamrei R, Ghorbanian A. Topical diltiazem vs. topical glyceril trinitrate in the treatment of chronic anal fissure: a prospective, randomized, double-blind trial. Acta Gastroenterol Belg. 2012 Dec;75(4):438-42. PMID 23402088
- [Result] Cevik M, Boleken ME, Koruk I, Ocal S, Balcioglu ME, Aydinoglu A, Karadag CA. A prospective, randomized, double-blind study comparing the efficacy of diltiazem, glyceryl trinitrate, and lidocaine for the treatment of anal fissure in children. Pediatr Surg Int. 2012 Apr;28(4):411-6. doi: 10.1007/s00383-011-3048-4. Epub 2012 Jan 3. PMID 22212494
- [Result] Kenny SE, Irvine T, Driver CP, Nunn AT, Losty PD, Jones MO, Turnock RR, Lamont GL, Lloyd DA. Double blind randomised controlled trial of topical glyceryl trinitrate in anal fissure. Arch Dis Child. 2001 Nov;85(5):404-7. doi: 10.1136/adc.85.5.404. PMID 11668104
- [Result] Tander B, Guven A, Demirbag S, Ozkan Y, Ozturk H, Cetinkursun S. A prospective, randomized, double-blind, placebo-controlled trial of glyceryl-trinitrate ointment in the treatment of children with anal fissure. J Pediatr Surg. 1999 Dec;34(12):1810-2. doi: 10.1016/s0022-3468(99)90318-4. PMID 10626860
- [Result] Nelson RL, Thomas K, Morgan J, Jones A. Non surgical therapy for anal fissure. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD003431. doi: 10.1002/14651858.CD003431.pub3. PMID 22336789
- [Result] Gremse DA, Hixon J, Crutchfield A. Comparison of polyethylene glycol 3350 and lactulose for treatment of chronic constipation in children. Clin Pediatr (Phila). 2002 May;41(4):225-9. doi: 10.1177/000992280204100405. PMID 12041718
- [Result] Dupont C, Leluyer B, Maamri N, Morali A, Joye JP, Fiorini JM, Abdelatif A, Baranes C, Benoit S, Benssoussan A, Boussioux JL, Boyer P, Brunet E, Delorme J, Francois-Cecchin S, Gottrand F, Grassart M, Hadji S, Kalidjian A, Languepin J, Leissler C, Lejay D, Livon D, Lopez JP, Mougenot JF, Risse JC, Rizk C, Roumaneix D, Schirrer J, Thoron B, Kalach N. Double-blind randomized evaluation of clinical and biological tolerance of polyethylene glycol 4000 versus lactulose in constipated children. J Pediatr Gastroenterol Nutr. 2005 Nov;41(5):625-33. doi: 10.1097/01.mpg.0000181188.01887.78. PMID 16254521
- [Result] Voskuijl W, de Lorijn F, Verwijs W, Hogeman P, Heijmans J, Makel W, Taminiau J, Benninga M. PEG 3350 (Transipeg) versus lactulose in the treatment of childhood functional constipation: a double blind, randomised, controlled, multicentre trial. Gut. 2004 Nov;53(11):1590-4. doi: 10.1136/gut.2004.043620. PMID 15479678
- [Result] Carapeti EA, Kamm MA, Phillips RK. Topical diltiazem and bethanechol decrease anal sphincter pressure and heal anal fissures without side effects. Dis Colon Rectum. 2000 Oct;43(10):1359-62. doi: 10.1007/BF02236630. PMID 11052511